CLINICAL TRIAL: NCT00333814
Title: A Study of the Safety and Efficacy of a New Treatment for Non-Infectious Intermediate or Posterior Uveitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206207-014
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-03

CONDITIONS: Intermediate Uveitis; Posterior Uveitis
MeSH Terms: conditions — Uveitis, Intermediate; Uveitis, Posterior | interventions — Dexamethasone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): Dexamethasone 350 µg
  Interventions: Drug: Dexamethasone
- 2 (Active Comparator): Dexamethasone 700 µg
  Interventions: Drug: dexamethasone
- 3 (Sham Comparator): Sham
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 350 µg; injection drug delivery system at Day 0
  Other Names: Posurdex®
  Arms: 1
Drug: dexamethasone — Dexamethasone 700 µg injection drug delivery system at Day 0
  Other Names: Posurdex®
  Arms: 2
Drug: Sham injection — Sham injection at Day 0
  Arms: 3

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone for the treatment of non-infectious intermediate or posterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with a diagnosis of chronic intermediate uveitis in at least one eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Any active ocular infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (18):
- Dallas, Texas, United States
- Sydney, Australia
- Vienna, Austria
- São Paulo, São Paulo/SP, Brazil
- Montreal, Quebec, Canada
- Prague, Czechia
- Paris, France
- Heidelberg, Germany
- Cholargós, Greece
- Hyderabad, India
- Petah Tikva, Israel
- Gdansk, Poland
- Coimbra, Portugal
- Johannesburg, South Africa
- Seoul, South Korea
- Madrid, Spain
- Lausanne, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Lightman S, Belfort R Jr, Naik RK, Lowder C, Foster CS, Rentz AM, Cui H, Whitcup SM, Kowalski JW, Revicki DA. Vision-related functioning outcomes of dexamethasone intravitreal implant in noninfectious intermediate or posterior uveitis. Invest Ophthalmol Vis Sci. 2013 Jul 18;54(7):4864-70. doi: 10.1167/iovs.12-10981. PMID 23761087
- [Derived] Naik RK, Rentz AM, Foster CS, Lightman S, Belfort R Jr, Lowder C, Whitcup SM, Kowalski JW, Revicki DA. Normative comparison of patient-reported outcomes in patients with noninfectious uveitis. JAMA Ophthalmol. 2013 Feb;131(2):219-25. doi: 10.1001/2013.jamaophthalmol.102. PMID 23411886
- [Derived] Lowder C, Belfort R Jr, Lightman S, Foster CS, Robinson MR, Schiffman RM, Li XY, Cui H, Whitcup SM; Ozurdex HURON Study Group. Dexamethasone intravitreal implant for noninfectious intermediate or posterior uveitis. Arch Ophthalmol. 2011 May;129(5):545-53. doi: 10.1001/archophthalmol.2010.339. Epub 2011 Jan 10. PMID 21220619
- See also: Related Info — http://www.allerganclinicaltrials.com/inquiries/trialsubject.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone 350 µg: Dexamethasone 350 µg
- Dexamethasone 700 µg: Dexamethasone 700 µg
- Sham: Sham
Period: Overall Study
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham
Started | 76 | 77 | 76
Completed | 73 | 73 | 71
Not Completed | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham | Total
Number analyzed (Participants) | 76 | 77 | 76 | 229
Age, Customized [Number; unit: Participants]
  <45 years | 39 | 43 | 41 | 123
  Between 45 and 65 years | 32 | 28 | 27 | 87
  >65 years | 5 | 6 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 51 | 145
  Male | 28 | 31 | 25 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Vitreous Haze (Ocular Inflammation) Score of Zero
Description: Percentage of patients with Vitreous Haze Score of Zero at Week 8. Score is based on standardized scale of 0 to +4 where 0 equals no inflammation and +4 equals optic nerve head not visible (severe).
Time Frame: Week 8
Population: Intent to Treat
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham
Number analyzed (Participants) | 76 | 77 | 76
Percentage of Patients | 35.5 | 46.8 | 11.8

2. Other Pre Specified Outcome: Percentage of Patients With at Least a 15-Letter Improvement in Best Corrected Visual Acuity (BCVA)
Description: Percentage of Patients with at least a 15-letter improvement in BCVA at Week 8 from Baseline. BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). An improvement in the number of letters read means that the vision has improved.
Time Frame: Week 8
Population: Intent to Treat
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham
Number analyzed (Participants) | 76 | 77 | 76
Percentage of Patients | 39.5 | 42.9 | 6.6

3. Other Pre Specified Outcome: Percentage of Patients With at Least a 10-Point Improvement in the National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25)Score
Description: Percentage of patients with at least a 10-Point Improvement in the NEI-VFQ-25 over-all composite score at Week 8 from Baseline. The NEI-VFQ-25 consists of 25 vision-targeted questions plus one general health question resulting in a score of 0-100 (100 represents best functionality).
Time Frame: Week 8
Population: Intent to Treat
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham
Number analyzed (Participants) | 76 | 77 | 76
Percentage of Patients | 40.8 | 50.7 | 15.9

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated. The Intent-to-Treat population was used for the outcome measure analyses and is calculated as the number of patients that were randomized (or started the study).
Arm/Group | Dexamethasone 350 µg | Dexamethasone 700 µg | Sham
Serious Adverse Events (participants affected / at risk) | 6/74 | 7/76 | 5/75
Other Adverse Events (participants affected / at risk) | 58/74 | 61/76 | 51/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 350 µg (N=74) | Dexamethasone 700 µg (N=76) | Sham (N=75)
Retinal Detachment (Eye disorders) | 0 | 2 | 2
Endophthalmitis (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Necrotising retinitis (Eye disorders) | 1 | 0 | 0
Pupillary disorder (Eye disorders) | 1 | 0 | 0
Hypotony of eye (Eye disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
HIV test positive (Investigations) | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 350 µg (N=74) | Dexamethasone 700 µg (N=76) | Sham (N=75)
Conjunctival haemorrhage (Eye disorders) | 13 | 23 | 16
Intraocular pressure increased (Investigations) | 17 | 19 | 5
Eye Pain (Eye disorders) | 8 | 11 | 10
Iridocyclitis (Eye disorders) | 2 | 11 | 5
Uveitis (Eye disorders) | 7 | 10 | 10
Ocular discomfort (Eye disorders) | 3 | 10 | 6
Cataract (Eye disorders) | 6 | 9 | 7
Myodesopsia (Eye disorders) | 5 | 7 | 5
Ocular hypertension (Eye disorders) | 7 | 6 | 0
Conjunctival hyperaemia (Eye disorders) | 7 | 5 | 7
Headache (Nervous system disorders) | 6 | 5 | 5
Vision blurred (Eye disorders) | 4 | 5 | 3
Eye irritation (Eye disorders) | 2 | 4 | 3
Intermediate uveitis (Eye disorders) | 0 | 4 | 1
Visual acuity reduced (Eye disorders) | 7 | 3 | 6
Macular oedema (Eye disorders) | 4 | 3 | 6
Eye pruritis (Eye disorders) | 3 | 3 | 5
Cataract subcapsular (Eye disorders) | 5 | 2 | 4
Conjunctivitis (Eye disorders) | 3 | 1 | 4
Eye swelling (Eye disorders) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.